CLINICAL TRIAL: NCT07272967
Title: Safety and Efficacy of Metformin in Preventing Secondary Gliosis Following Acute Thoraco-Lumbar Spinal Cord Injury: A Randomized, Double-Blinded, Placebo-Controlled Study.
Brief Title: Metformin in Preventing Secondary Gliosis Following Acute Thoraco-Lumbar Spinal Cord Injury
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Badr University (Other)
Responsible Party: Principal Investigator, Eman Said Sawan, Lecturer of Clinical Pharmacy, Faculty of Pharmacy, Badr University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 9/2025NEUS6
Record Dates: First submitted 2025-11-19; First posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-11

CONDITIONS: Spinal Cord Injury (SCI)
Keywords: Metformin; spinal cord injury,; gliosis; , randomized controlled trial; neuroprotection
MeSH Terms: conditions — Spinal Cord Injuries; Gliosis | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Metformin (Active Comparator): The metformin group will receive 1,000 mg of immediate-release metformin orally, twice daily
  Interventions: Drug: Metformin
- Placebo (Placebo Comparator): Participants in the placebo group will receive an identical-appearing placebo, administered orally, twice daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Metformin — Participants assigned to the metformin group will receive 1,000 mg of immediate-release metformin orally, twice daily
  Other Names: Glucophage 1000 mg tablets
  Arms: Metformin
Drug: Placebo — Participants in the placebo group will receive an identical-appearing placebo, administered orally, twice daily
  Other Names: Metformin free tablets
  Arms: Placebo

SUMMARY:
Background:

Spinal cord injury (SCI) is a major global health problem, with thoraco-lumbar injuries often leading to paraplegia and incomplete neurological recovery. The glial scar, resulting from astrocyte activation at the injury site, constitutes a major barrier to axon regeneration. Given the limitations of current treatments, there is an urgent need for new interventions to improve outcomes. Metformin, a common drug for diabetes, shows promising potential as a neuroprotective agent in preclinical SCI models, where it improves motor function and reduces pain and glial scar formation. Its safety in acute neurological injury has also been supported in a recent human trial for severe traumatic brain injury.

Objective:

To test the safety and efficacy of metformin in acute thoraco-lumbar SCI, focusing on neurological and functional outcomes as well as DTI metrics of spinal cord integrity.

Methods. Study Design. Randomized, double-blinded, placebo-controlled study.

Population:

Participants that will be admitted during the time of the study to Neurosurgery department at Menoufia University hospitals at Menoufia University.

Setting:

Neurosurgery department at Menoufia University hospitals at Menoufia University.

Keywords:

Metformin, spinal cord injury, gliosis, randomized controlled trial, neuroprotection

DETAILED DESCRIPTION:
Study Design. Randomized, double-blinded, placebo-controlled study. Randomization and Blinding. Participants will be randomly assigned to either the metformin or placebo group in a 1:1 ratio using block randomization. A computer-generated randomization sequence will be created with the R software (version 4.4.1) and the blockrand package(7). This sequence will be securely stored and accessible only to the study statistician. Treatment packets will be pre-labeled with unique numbers matching the randomization sequence. When a patient qualifies for the study, they will receive a numbered packet corresponding to their assignment. To ensure objectivity, neither participants nor study staff will know which number corresponds to metformin or placebo-only the statistician will have access to this information.

Setting:

Neurosurgery department at Menoufia University hospitals at Menoufia University.

Instruments:

We will assess the patient using AISA grade, Visual Analog Scale (VAS) and the Neuropathic Pain Symptom Inventory (NPSI) (8-10).

Data collection:

It will be done by data collaborators under the leadership of the investigators in: Neurosurgery department at Menoufia University hospitals at Menoufia University.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-65 years, who had acute, non-penetrating thoraco-lumbar SCI (T1-conus medullaris), with new neurological deficits.
* Injury occurred within the past 24 hours before enrollment.
* American Spinal Injury Association (ASIA) Impairment Scale grade B-D.
* Able to undergo MRI of the spine.
* Informed consent provided by patient or legal representative.

Exclusion Criteria:

* Major spinal transaction or cervical spinal cord injury.
* Prior spinal surgery or pre-existing spinal pathology (e.g., kyphosis, tumors).
* Concomitant severe traumatic brain injury (Glasgow Coma Scale < 13) or other CNS injury that would confound neurological assessment.
* Known diabetes mellitus (type 1 or 2) or current use of metformin.
* Penetrating spinal injury (e.g. gunshot, stab wound).
* Implanted metallic devices or conditions precluding MRI.
* Pregnancy or breastfeeding.
* Severe comorbidities (e.g. end-stage liver disease, renal failure with eGFR<30 mL/min).
* Known allergy to metformin.
* Uncontrolled infection or sepsis at presentation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Neurological recovery | 2 weeks, and 3-months postoperatively.
  Comparison of postoperative American Spinal Injury Association (ASIA) Impairment Scale grade ranging from A to E where Grade A= Complete spinal cord injury and Grade E=Normal function

SECONDARY OUTCOMES:
Pain intensity | at 2 weeks, and 3-months postoperatively
  Comparison of postoperative patient-reported pain using Visual Analog Scale (VAS) that is ranging from 0-10 score where 0=no pain and10= the worst possible pain
Neuropathic Pain character | at 2 weeks, and 3-months postoperatively
  Comparison of postoperative Neuropathic character of pain using Neuropathic Pain Symptom Inventory (NPSI) scale ranging from 0-10 score where 0=no pain and 10= the worst possible pain

CONTACTS AND LOCATIONS:
Locations (1):
- Neurosurgery department at Menoufia University hospitals at Menoufia University., Shibīn al Kawm, Menoufia, Egypt

IPD SHARING:
Plan to Share IPD: No
Data is available with corresponding author on reasonable request